CLINICAL TRIAL: NCT05961475
Title: Evaluating the Postprandial Glucose Response After Fruit Snack Consumption
Brief Title: Monitoring Postprandial Glycemia in Fruit Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean Spray Cranberries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BIO-2309
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First product order: order not stated to protect study blinding (Experimental): Participants will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit Snack 2; Dietary Supplement: Fruit Snack 3; Dietary Supplement: Fruit Snack 4; Dietary Supplement: White Bread
- Second product order: order not stated to protect study blinding (Experimental): Participants will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit Snack 2; Dietary Supplement: Fruit Snack 3; Dietary Supplement: Fruit Snack 4; Dietary Supplement: White Bread
- Third product order: order not stated to protect study blinding (Experimental): Participants will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit Snack 2; Dietary Supplement: Fruit Snack 3; Dietary Supplement: Fruit Snack 4; Dietary Supplement: White Bread
- Fourth product order: order not stated to protect study blinding (Experimental): Participants will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit Snack 2; Dietary Supplement: Fruit Snack 3; Dietary Supplement: Fruit Snack 4; Dietary Supplement: White Bread
- Fifth product order: order not stated to protect study blinding (Experimental): Participants will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit Snack 2; Dietary Supplement: Fruit Snack 3; Dietary Supplement: Fruit Snack 4; Dietary Supplement: White Bread

INTERVENTIONS:
Dietary Supplement: Fruit snack 1 — Fruit snacks with original level of sugar
Dietary Supplement: Fruit Snack 2 — Fruit snacks with original level of sugar and mulberry leaf extract
Dietary Supplement: Fruit Snack 3 — Fruit snacks with reduced level of sugar
Dietary Supplement: Fruit Snack 4 — Fruit snacks with zero added sugar
Dietary Supplement: White Bread — White bread with matched carbohydrate as control

SUMMARY:
The goal of this clinical trial is to compare the postprandial glucose and insulin responses after different fruit snack consumption in a healthy population.

DETAILED DESCRIPTION:
Fruit snacks made from sweetened dried fruits is a source of polyphenols, fiber, and other nutrients. The addition of sugar could aid in the taste, texture, and shelf life of these types of products. Fruit snacks with different levels of sugar were developed to meet various consumer needs. The postprandial glucose response in a healthy population is of interest in this regard.

Mulberry leaf extract has been shown the benefit of blood glucose regulation in multiple studies. This is mainly due to the function of the most predominant iminosugar, 1-deoxynojirimycin (DNJ), in the mulberry leaf extract which acts as α-glucosidase inhibitor. Fruit snacks containing mulberry leaf extract were developed and the postprandial metabolic response against a reference (white bread matched for carbohydrate) will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 to ≤45 years of age at visit 1.
2. BMI ≥18.5 and <30.0 kg/m2 at visit 1.
3. Fasting capillary glucose <100 mg/dL at visit 1.
4. Willing to avoid consuming high-polyphenol containing foods (Appendix 2) for 48 h prior to each test visit.
5. Willing to abstain from alcohol consumption for 24 hours prior to each study visit.
6. Non-user of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1, with no plans to begin use during the study period.
7. Willing to maintain habitual physical activity level throughout the duration of the study.
8. Willing to maintain habitual dietary pattern throughout the duration of the study, including stable intake of current vitamins, minerals, supplements and medications not interfering with study outcomes.
9. Score of 7 to 10 on the Vein Access Scale at visit 1 (Appendix provided for further checking).
10. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
11. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurological disorders that may affect the subject's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
2. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit 1 (3 repeated measurements will be taken after subjects sit quietly for at least 5 mins. Each measurement will be separated by at least 2 minutes. The average of the last two measurements will be used).
3. Unstable use (initiation or change in dose) within 30 days of visit 1 of antihypertensive medications.
4. Unstable use (initiation or change in dose) within 30 days of visit 1 of thyroid hormone replacement medications.
5. Use of medications or supplements that may influence carbohydrate metabolism within 30 days of visit 1.
6. Extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian) at the discretion of the Clinical Investigator.
7. Weight loss or gain >4.5 kg in the 2 months prior to visit 1.
8. Currently, or planning to be, on a weight loss regimen during the study.
9. Use of weight loss medication within 90 d of visit 1.
10. History of gastrointestinal surgery for weight reducing purposes.
11. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
12. Known allergy or sensitivity to any ingredients or potential allergens contained in the study product.
13. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
14. History of any major trauma or major surgical event within 2 months of visit 1.
15. Blood donation >450 mL within 8 weeks of visit 2 or plans to donate blood or plasma during the study period.
16. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential with unstable use (initiation or change in dose) within 30 days of visit 1) of sex hormones for contraception.
17. Recent history of (within 12 months of screening; visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
18. Exposed to any non-registered drug product within 30 days prior to visit 1.
19. Any condition the Investigator believes would interfere with the subject's ability to provide informed consent or comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Glucose maximal concentration (Cmax) 2 hours after consumption | 2 hour after consumption
  Glucose Cmax

SECONDARY OUTCOMES:
Glucose incremental area under the curve (iAUC) from pre-product consumption to 120 min | 2 hours
  Glucose iAUC
Glucose time to maximum concentration within 2 hours after consumption | 2 hours
  Glucose Tmax
Insulin incremental area under the curve (iAUC) from pre-product consumption to 120 min | 2 hours
  Insulin iAUC
Insulin maximal concentration (Cmax) 2 hours after consumption | 2 hours
  Insulin Cmax
Insulin time to maximum concentration within 2 hours after consumption | 2 hours
  Insulin Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No